CLINICAL TRIAL: NCT07320651
Title: Improving Shared Decision-Making in Menstrual Management and Contraception for Adolescents and Young Adults: A Cluster-Randomized Trial
Brief Title: Improving Shared Decision-Making in Menstrual Management and Contraception for Adolescents and Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Dehlia Moussaoui, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-00733
Record Dates: First submitted 2025-08-31; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Contraception; Menstrual Management
Keywords: decision aid; menstrual management; contraception; shared decision-making

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Other: Standard counseling
- intervention group (Experimental)
  Interventions: Other: Encounter decision aid

INTERVENTIONS:
Other: Encounter decision aid — The intervention will involve the use of an encounter decision aid (EDA) during the clinical encounter. This paper-based tool was developed through an iterative process at HUG by our multidisciplinary team, comprising clinicians, specialized nurses, clinical researchers, graphic designer, stakeholders and patient representatives.
  Arms: intervention group
Other: Standard counseling — The control intervention consists of standard consultation with usual counseling.
  Arms: control group

SUMMARY:
Decision aids are educational tools designed to help people participate in decision-making about health care choices, by providing evidence-based information, promoting patient-centered care, and supporting patient autonomy and engagement. Our research team developed an Encounter Decision Aid (EDA) exploring treatment options for menstrual management in adolescents and young adults (AYAs), in accordance with the latest International Patient Decision Aids Standards and the Ottawa Decision Support Framework.

In this cluster-randomized controlled trial, we aim to evaluate the effectiveness of this EDA on patient-centered outcome measures in AYAs considering treatment for menstrual management and/or contraception compared to standard counseling.

ELIGIBILITY:
Inclusion Criteria:

* adolescents and young adults aged 12-25 years old
* presenting to an outpatient consultation at "Unité de policlinique de gynécologie" or "Consultation de gynécologie pédiatrique" at HUG
* considering initiation or switch to hormonal medication for menstrual management and/or contraception
* able to give informed consent as documented by signature or accompanied by a legal guardian who can provide consent if required.

Exclusion Criteria:

* individuals who cannot read and understand French to a degree that would prevent participation in informed consent and study-related materials.
* individuals who have major sensory disability, such as visual or hearing impairment, that would compromise their ability to give written informed consent and use the EDA, in the absence of their legal guardian.
* individuals with cognitive or psychiatric conditions significantly impairing decision making capacity, unless accompanied by a legal guardian.
* patients currently participating in another clinical trial related to contraceptive decision-making, to avoid potential interference.

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Patient decisional conflict measured using the Decisional Conflict Scale low literacy (LL-DCS). | immediately after the clinical encounter
  Decisional conflict is defined as a state of uncertainty about a course of action and is measured by the Decisional Conflict Scale. It is recognized as a core component of the quality of the decision-making process. The Decisional Conflict Scale low literacy (LL-DCS) is a validated score that includes 10 items which are scored on a 0 to 4 scale; the items scores are summed, divided by 10, and then multiplied by 25. The total score ranges from 0 to 100, with higher scores indicating greater decisional conflict.

SECONDARY OUTCOMES:
Patient decisional conflict at 3 months, using the low literacy Decisional Conflict Scale (LL-DCS). | at 3 months post-clinical encounter
  Decisional conflict is defined as a state of uncertainty about a course of action and is measured by the Decisional Conflict Scale. It is recognized as a core component of the quality of the decision-making process. The Decisional Conflict Scale low literacy (LL-DCS) is a validated score that includes 10 items which are scored on a 0 to 4 scale; the items scores are summed, divided by 10, and then multiplied by 25. The total score ranges from 0 to 100, with higher scores indicating greater decisional conflict.
Patient knowledge. | immediately after the clinical encounter
  Score on a 7-item true/false questionnaire on hormonal treatment and contraception, assessed right after the clinical encounter.
Knowledge retention | knowledge questionnaire at 3 months post-intervention
  Reassessment of knowledge using the same questionnaire (score on a 7-item true/false questionnaire on hormonal treatment and contraception) at 3 month-follow up.
Patient and healthcare provider satisfaction with the decision-making process | immediately after the clinical encounter
  * Patient satisfaction rated on a 5-point Likert scale, indicating how strongly they would recommend the decision-making approach.
  * Clinician satisfaction rated on a 5-point Likert scale (where higher scores indicating greater satisfaction). Satisfaction will be defined as the proportion scoring ≥4 ("very satisfied" and extremely satisfied").
Patient involvement in decision-making | immediately after the clinical encounter (10-point Likert scale).
  measured by the self-reported collaboRATE scale (three brief questions that patients complete following the clinical encounter)
Patient involvement in decision-making | immediately after the clinical encounter
  assessed via the OPTION-5 instrument (where independent observer rate clinician behaviors on a standardized scale (0-100), applied to a video recording of the clinical encounter).
Participant treatment preference before the clinical encounter | Baseline
  self-reported answer to the question: "Which treatment would you like to start?"
Participant treatment preference after the clinical encounter | Immediately after the clinical encounter
  self-reported answer to the question: "Which treatment would you like to start?"
Medication continuation | at 3 months
  self-reported answer to the question: "if a medication was prescribed following your previous gynecological appointment, are you still currently using it?" yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided